CLINICAL TRIAL: NCT02882737
Title: The Impact of Subcutaneous Glucagon Before, During and After Exercise a Study in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Isabelle Steineck, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 16016762
Record Dates: First submitted 2016-08-17; First posted 2016-08-30 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2016-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise and glucagon before exercise (Experimental): 120 minutes after breakfast; a single subcutaneous bolus of 200µg glucagon is administered by the primary investigator. However, the patient do, not know whether placebo or a glucagon injection is administered.
  Exercise: Immediately thereafter, the patient will bicycle for 45 minutes at 50% of the heart rate HR reserve.
  When exercise is ended a single subcutaneous bolus of 0.2 ml saline is administered and the exercise session will be suspended. Again, the patient do not know whether placebo or a glucagon is administered.
  Interventions: Drug: Glucagon before exercise
- Exercise and glucagon after exercise (Active Comparator): 120 minutes after breakfast; a single subcutaneous bolus of 0.2 ml saline is administered by the primary investigator. However, the patient do, not know whether placebo or a glucagon injection is administered.
  Exercise: Immediately thereafter, the patient will bicycle for 45 minutes at 50% of the heart rate HR reserve.
  Low-dose glucagon phase: When exercise is ended or when hypoglycemia occurs (≤3.9 mmol/l); a single subcutaneous bolus of 200μg glucagon is administered and the exercise session will be suspended. Again, the patient do not know whether placebo or a glucagon is administered.
  Interventions: Drug: Glucagon after exercise
- Resting and glucagon after resting (Active Comparator): 120 minutes after breakfast; a single subcutaneous bolus of 200μg placebo is administered.
  Resting: After placebo injection the patient will be resting on a hospital bed for 45 minutes. The patient do not know if placebo or glucagon is administered.
  Low-dose glucagon phase: After 45 minutes of resting or when hypoglycemia occurs, a single subcutaneous bolus of 200μg glucagon is administered.
  Safety issues: If plasma glucose drops < 2.5 mmol/l at two consecutive measurements with 5 min interval or the patient experiences unbearable symptoms of hypoglycemia even after glucagon administration, 20 g carbohydrate is given orally. If plasma glucose drops< 2.3 mmol/l or doesn't raise sufficient after oral glucose, we will give intravenøs glucose to the patient. The study will then end and a new study day will be planned.
  Interventions: Drug: Glucagon after resting

INTERVENTIONS:
Drug: Glucagon before exercise
  Arms: Exercise and glucagon before exercise
Drug: Glucagon after exercise
  Arms: Exercise and glucagon after exercise
Drug: Glucagon after resting
  Arms: Resting and glucagon after resting

SUMMARY:
This project is part of several studies exploring situations, where glucagon potential has lesser glucose elevating effect. Exercise can be one of these situations as exercise may reduce liver glycogen depots.

The investigators aims are:

1. To compare the increase in plasma glucose after 200µg glucagon given either after exercise or after resting for 45 minutes.
2. To determine whether a subcutaneous glucagon injection just before exercise has a greater impact on hepatic glucose production and thereby is superior to an injection after exercise in preventing hypoglycemia during and two hours after exercise.
3. To compare the accuracy of two Dexcom G4 continuous glucose monitors, (CGM) placed at either the abdominal wall or on the upper arm.

DETAILED DESCRIPTION:
Design:

A randomized placebo-controlled single-blinded study will be conducted. The subjects do not know if they get glucagon or placebo but the investigator know if the subject get glucagon or placebo. Study participants have to complete three study days and serve as their own controls. After participants have given an informed consent, they will go through three steps:

1. Screening day
2. Run-in period
3. Three study days in a random order:

   * Exercise and glucagon injected after cycling/or during cycling in case of hypoglycemia
   * Resting and glucagon after resting
   * Exercise and glucagon subcutaneous before cycling

47-49 hours before the study visits one CGM device is placed on the abdominal wall on the participant at least 7 cm from the site of the insulin pump infusion set. One CGM is placed on the non-dominant upper arm between 10 cm from elbow and 10 cm from shoulder on the posterior/lateral side on the arm. The CGMs will be in place for seven days. The CGM readings on the CGM placed at the abdominal wall are not blinded for the participant. The CGM readings on the CGM placed on the arm is blinded for the participant. In the period from the study visits to 4 days after the study visits the participant will do self-monitoring of blood glucose 8 times a day on standardized times.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes ≥ 2 year
* BMI 20-30 kg/m2
* Insulin pump ≥ 1 year.
* HbA1c < 69 mmol/mol (8.5 %)
* Hypoglycemia awareness (reported by Gold et al.)
* Use of carbohydrate counting and the insulin pump bolus calculator for all meals
* Sedentary or mild physical activity: Less than 150 minutes of moderate-intensity aerobic physical activity throughout the week and less than 75 minutes of vigorous-intensity aerobic physical activity throughout the week .

Exclusion Criteria:

* Allergy or intolerance to lactose or GlucaGen® (Novo Nordisk, Bagsværd, DK)
* Impaired renal function (eGFR < 60 ml/min/1.73m2)
* Liver disease with ALAT > 2.5 times the upper limit of the reference interval
* Use of anti-diabetic medicine (other than insulin), per oral corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start
* Known or suspected alcohol or drug abuse
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation
* Females who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods
* Inability to understand the patient information and to give informed consent
* Physical or mental incapacity to perform exercise
* Chronic use or unable to stop acetaminophen (paracetamol) use
* Allergy to the patch of CGM

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is peak plasma glucose achieved within 2 hours after the 200 μg subcutaneous glucagon injection. In the primary analysis, the investigators will compare the peak plasma glucose after exercise and after resting. | 2 hours

SECONDARY OUTCOMES:
The time-to-peak value after glucagon injection. | 2 hours
Duration of the glucagon effect; equal to the time point from glucagon injection to when plasma glucose is below baseline. | 2 hours
The glycaemic effect, calculated as the total area under the curve (tAUC) after each glucagon injection. | 2 hours
Changes in plasma ketone bodies after each glucagon injection. | 2 hours
Changes in plasma lactic acid after each glucagon injection | 2 hours
Changes in plasma glucagon after each glucagon injection | 2 hours
Changes in serum free fatty acid (FFA) after each glucagon injection | 2 hours
Changes in serum triglycerides after each glucagon injection | 2 hours
Number of events of hypoglycemia (plasma glucose ≤3.9 mmol/l) in the three study days. | 3 hours
Number of re-events of hypoglycemia (plasma glucose ≤3.9 mmol/l) 30 minutes after first event in the three study groups. | 30 minutes
Number of rebound hyperglycemia (plasma glucose ≥10.0 mmol/l). | 4 hours
Mean absolute difference (MARD) in the two CGM sites during the four days after the study day using the daily 8 prespecified plasma glucose measurements by Bayer Contour Link as the reference value. | 4 days
Mean absolute relative difference (MARD) during the study visits between the two sensor sites with the YSI 2300 STAT PLUS as the reference value. | 6 hours
MARD during the hypoglycemia range (≤3.9 mmol/l) of the study visits between the two sensor sites (CGMarm vs. CGMabdomen) with the YSI 2300 STAT PLUS as the reference value. | 6 hours
MARD during the euglycemia range (>3.9 mmol/l and < 10.0 mmol/l) of the study visits between the two sensor sites (CGMarm vs. CGMabdomen) with the YSI 2300 STAT PLUS as the reference. | 6 hours
MARD during the hyperglycemia range (≥10.0 mmol/l) of the study visits for the two Dexcom G4 sensor sites (CGMarm vs. CGMabdomen) with the YSI 2300 STAT PLUS as the reference value | 6 hours
MARD for the two sensor sites (CGMarm and CGMabdomen) from day 1- 7 with the Bayer Contour Link as the reference value. | 7 days
The rate-of change (ROC) of the two sensors. | 6 hours
The rate-of change (ROC) of plasma glucose measured by the YSI 2300 STAT PLUS. | 6 hours
The Precision Absolute Relative Difference (=CGM readings of one system will be subtracted from CGM readings of the other system, and this difference will be divided by the average of the CGM readings of the abdominal sensors.) | 7 days
The sensors' sensitivity and specificity to detect a hypoglycemic event. | 7 days
The point accuracy of both sensors with the Clarke error grid analysis | 7 days
The pressure induced sensor attenuation (PISA) by using a recent fault detection algorithm that can detect non-physiologic anomalous low sensor readings. | 7 days
The fused data from the two sensors. | 7 days
  Fused data will be compared with data from individual sensors

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Steineck, MD, Principal Investigator — Hvidovre Hospital department of endocrinology
Locations (1):
- Isabelle Steineck, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data are processed and merged into at least two scientific articles published in international peer-reviewed scientific journal. Positive, negative and inconclusive results will be published as soon as scientifically justifiable. The study protocol will be published at www.clinicaltrial.gov. The results from the study will within 1 year be published on EudraCT. The sponsor will contact the Danish Health and Medicines Authority within 90 days after the study is ended and to inform them that the study has ended

REFERENCES:
- [Derived] Steineck IIK, Ranjan A, Schmidt S, Clausen TR, Holst JJ, Norgaard K. Preserved glucose response to low-dose glucagon after exercise in insulin-pump-treated individuals with type 1 diabetes: a randomised crossover study. Diabetologia. 2019 Apr;62(4):582-592. doi: 10.1007/s00125-018-4807-8. Epub 2019 Jan 14. PMID 30643924